CLINICAL TRIAL: NCT06860685
Title: A Non-randomised External Controlled Trial of Gum Chewing to Enhance the Restoration of Intestinal Motility in Colorectal Surgery
Brief Title: Trial of Gum Chewing to Enhance the Restoration of Intestinal Motility in Colorectal Cancer Surgery
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Hui Yang, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SCCHEC-02-2020-059
Record Dates: First submitted 2025-02-21; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Chewing Gum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gum chewing in high-risk group (Experimental): Patients will receive enhanced recovery care and gum chewing (three times per day) on the first postoperative morning until oral dietary intake.
  Interventions: Dietary Supplement: gum chewing
- Control in low-risk group (No Intervention): Patients only receive Enhanced recovery care, including no administration of intestinal antibiotics; normal diet until 6 hours before surgery; no nasogastric drainage; minimal perioprative intravenous fluid; patient started to ambulate and drink water on the first postoperative day

INTERVENTIONS:
Dietary Supplement: gum chewing — Participants allocated to chewing gum will be instructed to chew commercially available sugar-free gum (Extra & Reg, Wm. Wrigley Jr. Co., Ltd., Shanghai, China) three times daily from the first postoperative morning until oral dietary intake. They were instructed to chew the piece of gum for at least 10 minutes.
  Arms: gum chewing in high-risk group

SUMMARY:
Surgery is one of the most frequent treatments of colorectal cancer. However, delayed restoration of intestinal motility is a common phenomenon in patients who undergo colorectal surgery, and may reduce comfort, prevent the early hospital discharge of patients and increase healthcare costs. Gum chewing is a kind of safe and easily accessible sham feeding to stimulate intestinal motility. In addition, prediction models were used to estimate the risk of delayed restoration of intestinal motility after colorectal surgery. Thus, this study is an External Controlled trial that will determine whether stratified application of gum chewing by risk prediction model will enhance restoration of intestinal motility and reduce healthcare costs in paitents undergoing open or laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
Background:

Identifying patients at high risk of delayed restoration of intestinal motility at an early stage and adopting individualized interventions is crucial. The risk prediction model can provide a highly accurate, individualized evidence-based risk estimation by identifying risk factors and creating a risk stratification system. In addition, gum chewing is a kind of sham feeding that has been reported to stimulate intestinal motility and emerged as a popular, simple, safe, effective method for enhancing restoration intestinal motility. Thus, this study combines risk prediction model and gum chewing, aiming to use pre- and intraoperative risk factors to predict the risk of delayed restoration of intestinal motility. After creating a risk stratification system, patients with colorectal surgery will be stratified to high-risk group or low-risk group of delayed restoration of intestinal motility.

Objective:

To compare the efficacy and economics of gum chewing in patients undergoing open or laparoscopic colorectal surgery after stratification by a risk prediction model.

Design:

This is a single-center, two-arm, prospective study and non-randomized external controlled trial.

Subjects:

Two hundred and ninety-two consecutive patients undergoing open or laparoscopic colorectal surgery will be recruited in experiment group, which includes high-risk group and low-risk group.

Interventions:

The low-risk group will only receive enhanced recovery care and the high-risk group will be instructed to chew gum as well as receive enhanced recovery care. The enhanced recovery care consists of no administration of intestinal antibiotics and normal diet until 6 hours before surgery; no nasogastric drainage and minimal perioperative introvenous fluid on the day of surgery; patients start to ambulate and drink water on the first postoperative day. Patients in high-risk group are instructed to chew the piece of sugar-free gum three times (at least 10 minutes) a day from the first postoperative morning until oral dietary intake.

Outcome measures:

The outcomes are first flatus time、first defecation time、Proportion of delayed restoration of intestinal motility、length of hospital stay. All the patients will be assisted to fill in "Patient Log" about the first flatus time and first defecation time after surgery until the oral dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed colorectal cancer
* Undergo open or laparoscopic colorectal surgery
* Able to give informed consent
* With normal verbal skills

Exclusion Criteria:

* Preoperative lower extremity dysfunction
* Dysphagia before surgery
* Patients who are discharged ,transferred to another hospital or die within 72
* hours after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
first flatus time | end of surgery to first passage of flatus, up to 3 days
  time to the passage of first flatus
first defecation time | end of surgery to first passage of defecation, up to 3 days
  time to the first defecation
proportion of delayed restoration of intestinal motility | up to 3 days
  The proportion of delayed restoration of intestinal motility will be caculated as the number of participants with delayed restoration of intestinal motility divided by the total number of participants enrolled in the study
length of hospital stay | up to 30 days (till successful discharge from secondary care to home, up to 30 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Clinical Research Center for Cancer, Sichuan Cancer Hospital & Institute, Sichuan Cancer Center, Afffliated Cancer Hospital of University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No